CLINICAL TRIAL: NCT05435716
Title: Efficacy and Safety Trial of C-wave™ Peripheral Lithoclasty Catheter System in Peripheral Arterial Angioplasty
Brief Title: Clinical Trial of C-Wave™ Peripheral Lithoclasty System Catheter System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suzhou Zhonghui Medical Technology Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YYS-2021-07-01
Record Dates: First submitted 2022-06-15; First posted 2022-06-28 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-06

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peripheral seismic catheterization system (IVL) + drug-coated balloon (DCB) and/or stent (Experimental)
  Interventions: Device: C-wave™ peripheral seismic waveguide system
- PTA + DRUG-coated balloon (DCB) and/or stent (Other)
  Interventions: Device: Peripheral vascular balloon dilatation catheter (PTA)

INTERVENTIONS:
Device: C-wave™ peripheral seismic waveguide system — In the experimental group, if the target lesions did not show flow-limiting dissection or severe elastic retraction, drug-coated balloon was subsequently performed after lumen preparation by peripheral seismic catheterization system (IVL). If there is limited flow dissection or severe elastic retraction, stent therapy is followed.
  Arms: Peripheral seismic catheterization system (IVL) + drug-coated balloon (DCB) and/or stent
Device: Peripheral vascular balloon dilatation catheter (PTA) — Subjects in the control group received balloon dilatation catheter in peripheral blood for lumen preparation, and if the target lesions did not show flow-limiting interlayer or severe elastic retraction, drug-coated balloon therapy was subsequently performed. If there is limited flow dissection or severe elastic retraction, stent therapy is followed.
  Arms: PTA + DRUG-coated balloon (DCB) and/or stent

SUMMARY:
To evaluate the efficacy and safety of peripheral shock catheter system in peripheral arterial angioplasty.This trial is a prospective, multicenter, open, randomized, parallel controlled and superior clinical trial. Select ≥3 hospitals with the qualification of national clinical trial institutions as clinical trial centers, and plan to enroll a total of 120 subjects. The ratio of subjects in the trial group and the control group is 1: 1 (60 in the trial group and 60 in the control group). This study mainly includes four stages: the screening (baseline) period (-14 ~0 days), the operation day (the day of treatment), the postoperative visit (0~7days ) and the 30-day follow-up (30 ±7days ).

ELIGIBILITY:
Inclusion Criteria:

1. Age of subject is greater than or equal to 18.
2. Rutherford Grade 2~5;
3. The resting ABI of target limb ≤0.90, or ≤0.75 after exercise;
4. Agree to participate in this study and sign informed consent;
5. Estimated life expectancy >1 year.
6. According to the diagnosis of medical institutions or participating researchers, peripheral arterial tubuloplasty (including peripheral seismic catheterization system or peripheral vascular balloon dilatation catheter for lumen preparation, and subsequent drug-coated balloon therapy or stent implantation; Angiographic Inclusion Criteria
7. Target lesion that is located in a native, de novo superficial femoral artery (SFA) or popliteal artery (popliteal artery extends to and ends proximal to the ostium of the anterior tibial artery).
8. The target vessel has not received any prior surgical intervention (within 3 months), including endovascular therapy and open surgery, and the stenosis rate ≥ 50% or occlusive lesions were assessed preoperatively;
9. The target vessels were 2-7.5 mm in diameter and had at least one normal subgenicular outflow artery (stenosis rate ≤50%).
10. If the stenosis rate of the target lesion is 50-99% and the lesion length is less than or equal to 260mm, the target lesion may be continuous or intermittent, or both. If the target lesions were chronic occlusive lesions, the length of occlusive lesions was ≤100mm, and the total length of lesions was ≤260mm;
11. The calcification degree is at least moderate, which is defined as the presence of calcification signs in the vessels of the target lesions under CTA or fluoroscopy, and the calcification conditions are 1) located on both sides of the target lesions, 2) if the length of the target lesions is less than 50mm, the length of the calcification lesions is at least 20mm; If the target lesion length ≥50mm and < 100mm, the calcification lesion length should be at least 50% of the target lesion. If the target lesion length is ≥100mm, the calcification lesion length should be greater than 50mm.
12. If there are signs of acute or chronic thrombus in the target blood vessels, the above conditions are met after routine clinical treatment.

Note: Patients with inflow tract and outflow tract that are qualified for inclusion in this study after routine clinical treatment can be included. cc

Exclusion Criteria:

1. The Rutherford rating is 0, 1 and 6;
2. Severe infection of target limb requiring antibiotics or planned amputation above the ankle;
3. Previous intra-arterial therapy or open surgery had been performed on the target limb (within 1 month);
4. Coagulation abnormalities are known to exist;
5. Coagulation abnormalities are known to exist;
6. A history of stroke or myocardial infarction within 60 days;
7. Subjects who have participated in clinical trials of other medical devices or drugs during the same period;
8. Women who are pregnant or breastfeeding;
9. Other conditions that the investigator considers inappropriate for clinical trial participation; Angiographic Exclusion criteria
10. in-stent restenosis
11. A highly tortuous artery;
12. The inflow vessels upstream of the target lesion area have other obvious vascular lesions that have not been successfully treated (stenosis rate > 50%);
13. There is an aneurysm in the target vessel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-08-05 (Actual); Primary Completion 2023-09-08 (Estimated); Study Completion 2023-09-08 (Estimated)

PRIMARY OUTCOMES:
Technical Success Rate, TSR | Peri-Procedural
  Procedural success rate is defined as the ratio of participants whose residual stenosis ≤30% without flow-limiting dissection (≥ grade D) prior to DCB or stenting

SECONDARY OUTCOMES:
Primary patency rate of target lesion | Immediately after the procedure、 30 days
  as freedom from clinically-driven target lesion revascularization (TLR) and freedom from restenosis determined by duplex ultrasound or angiogram or CTA greater than or equal to 50% stenosis.
new-onset Major Adverse Events (MAEs) | 30 days
  Need for emergency surgical revascularization of target limb Unplanned target limb major amputation (above the ankle) Symptomatic thrombus or distal emboli that require surgical, mechanical or pharmacologic means to improve flow and extend hospitalization Perforations that require an intervention, including bail-out stenting
Clinical Success ABI | 30 days
  Defined as ankle-brachial index ABI reported as change from baseline
Clinical Success Rutherford Category | 30 days
  Defined as Rutherford Category reported as change from baseline
Performance of Device | Peri-Procedural
  Performance of Device is composed of as Guidewire compatibility；Introducer sheath compatibility；visibility of the catheter 、emitter and marker；catheter connection；corssing ability of thecatheter
Intraoperative complication | Peri-Procedural
Device defect (for test group only) | Peri-Procedural
  Device defects refer to unreasonable risks that may endanger human health and life safety, such as label errors, quality problems, failures.

CONTACTS AND LOCATIONS:
Locations (1):
- C-waveTM peripheral seismic waveguide system, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No